CLINICAL TRIAL: NCT06918821
Title: Reducing Obesity Through Play: A Randomized Control Trial
Brief Title: Reducing Obesity Through Play Among Toddlers: Tiny Steps to Health (TSHS) Study
Acronym: TSHS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Tracey Ledoux, Associate Professor, University of Houston
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 4899; R01HD114793-01 (NIH)
Record Dates: First submitted 2025-03-19; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Childhood Obesity
Keywords: toddlers; diet; physical activity; parenting
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Toddler Parent Group (HTPG) (Active Comparator): Parents assigned to HTPG will receive 10 weekly classes (60-minutes), which will include instruction on nutrition and physical activity for toddlers from a health educator with group discussion.
  Interventions: Behavioral: Healthy Toddler Parent Group (HTPG)
- Usual Lifestyle (No Intervention): Parent-toddler dyads assigned to the no treatment group will continue their normal day to day routine for 10-weeks. After parents and toddlers have participated in all data collection timepoints, they will receive a 1-month membership to a health club.
- Families Understanding Nutrition and Physically Active Lifestyles (FUNPALs) Playgroup (Experimental): Parent-toddler dyads assigned to this group will have access to 10-weekly playgroup sessions (90-minutes each). During sessions, parents and their toddler (and siblings) will be led by 2 facilitators through physical activities, healthy snack time (includes preparation), child-directed playtime, singing, parent coaching, and yoga stretches.
  Interventions: Behavioral: Families Understanding Nutrition and Physically Active Lifestyles (FUNPALs) Playgroup

INTERVENTIONS:
Behavioral: Healthy Toddler Parent Group (HTPG) — Parent education class
  Arms: Healthy Toddler Parent Group (HTPG)
Behavioral: Families Understanding Nutrition and Physically Active Lifestyles (FUNPALs) Playgroup — Family playgroup
  Arms: Families Understanding Nutrition and Physically Active Lifestyles (FUNPALs) Playgroup

SUMMARY:
The purpose of this study is to test various ways to help toddlers develop healthy eating and activity behaviors. Parents and toddlers, who participate in this research will be randomly assigned to either 1) continue their lifestyle behaviors for 10-weeks and then receive a health club membership for 1-month, 2) attend a health promotion playgroup together for 10 weeks, or 3) to attend an educational class for parents while toddlers are in childcare for 10-weeks. Physical measures of toddlers (height, weight, dietary intake, activity) will be collected. Parent-report surveys with questions about parenting, toddler diet, toddler temperament, food security status, demographic qualities, and satisfaction with group assignment will be collected. Last, the interactions between parents and toddlers will be observed and assessed during short play tasks via Zoom. All measures will be collected immediately upon signing up for the study (week 0), 10-weeks later (post), and 24-weeks after signing up for the study.

DETAILED DESCRIPTION:
In this randomized control trial, 300 parent-toddler dyads will be recruited and randomly assigned to one of three groups for 10-weeks. Those dyads assigned to the usual lifestyle group will not make any changes and will maintain their normal behaviors. Dyads assigned to the Families Understanding Nutrition and Physically Activity Lifestyles (FUNPALs) Playgroup will be invited to attend weekly playgroup sessions together. For those assigned to the Healthy Toddler Parent Group, parents will attend weekly health education classes where toddler health behaviors will be discussed. At baseline (week 0), immediate follow up (week 10-11), and long term follow up (week 24) parent report, physical, and observational measures of diet, activity, parenting, child temperament, food insecurity status, and quality of life will be completed.

ELIGIBILITY:
Inclusion criteria:

* Parents: Primary custodian (i.e., legal guardian) of a toddler, >18 years, have regular and frequent access to internet, fluent in English.
* Toddlers: >/=18 and </=36 months of age, and walking.

Exclusion criteria include:

* Parents or toddlers who have mental or physical conditions that would prevent engagement in nutrition, physical activity, play, or instructional activities in a group setting or families unwilling to commit to the whole program (e.g., planning to move) will be excluded because participants may be randomly assigned to group interventions where engagement in these activities will be expected.

  * Parents who are not fluent in English will be excluded because this study was developed, and pilot tested on an English-speaking population. All study materials are in English, the interventions will be offered in English, and most of the surveys are not available or have been validated for non-English speaking audiences.
  * Parents who are not willing or able to participate in parent-toddler interaction assessments via Zoom will be excluded. This assessment is an important study variable.
* Parents who are not willing to be recorded will be excluded because all Families Understanding Nutrition and Physically Active LIfestyles (FUNPALs) Playgroup sessions will be recorded for facilitator supervision purposes, and the parent-toddler interaction assessments will be recorded for later coding.
* Only one toddler and one parent per family will be eligible, but all children and siblings within a household will be able to attend playgroups or childcare while parents are in Healthy Toddler Parent Group (HTPG) classes.
* Parents and toddlers who received 1 or more sessions of the FUNPALs Playgroup or the HTPG. This study will be running 1 cohort per quarter for 4 years, so it is possible that families may drop out and want to re-enroll in a later cohort or enroll when younger siblings are eligible. They will not be eligible. Also, we will invite families from the community participate in practice sessions of FUNPALs or HTPG to train the facilitators. These families will not be eligible to participate in the study.

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-05-17 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Weight Status | baseline (T1), 10-11 weeks after baseline (T2), and 24- weeks after baseline (T3)
  Weight-for-length (WFL) percentile for toddlers <24 months. Length and weight measures will each be taken two times and averaged. Trained research assistants will measure height to the nearest 0.1 cm using a recumbent height board for children <24 months. Weight will be measured to the nearest 0.1 kg using an electronic self-calibrating digital scale. For toddlers <24 months, weight for length (WFL) will be calculated. Sex- and age-standardized WFL will be determined from Centers for Disease Control and Prevention (CDC) growth charts. Age and gender corrected WFL will be used to categorize weight status groups: <5th percentile WFL will be considered underweight, 5th-84.99th percentile will be considered normal weight, >85 percentile will be considered overweight and >95 percentile will be considered obese per CDC guidelines.
Weight Status | baseline (T1), 10-11 weeks after baseline (T2), and 24- weeks after baseline (T3)
  Body mass index (BMI) percentile for toddlers >/= 24 months. Height and weight measures will each be taken two times and averaged. Trained research assistants will measure height to the nearest 0.1 cm using a portable stadiometer for children >/=24 months. Weight will be measured to the nearest 0.1 kg using an electronic self-calibrating digital scale. For toddlers >/=24 months, BMI will be calculated. Sex- and age-standardized BMI percentiles will be determined from Centers for Disease Control and Prevention (CDC) growth charts. Age and gender corrected BMI percentile ranks will be used to categorize weight status groups: <5th percentile BMI will be considered underweight, 5th-84.99th percentile will be considered normal weight, >85 percentile will be considered overweight and >95 percentile will be considered obese per CDC guidelines.

SECONDARY OUTCOMES:
Toddler Dietary Intake. | baseline (T1), 10-11 weeks after baseline (T2), and 24- weeks after baseline (T3)
  National Cancer Institute's (NCI's) Automated Self-Administered 24 hour dietary recall (ASA24)- Parents will be sent a link on 3 non-consecutive days via email and/or text within a 1-week period of time. The link will take them to a series of questions to assess what their child has eaten and drank in the last 24-hours. The ASA24 system provides a complete nutritional analysis of the diet including servings of food groups and amounts of micro and macronutrients consumed. The average number of servings of fruits, vegetables, and whole grain foods; grams of sugar; and grams of saturated fat will be retained for this study.
Toddler carotenoid (FV) intake. | baseline (T1), 10-11 weeks after baseline (T2), and 24- weeks after baseline (T3)
  Child fruit and vegetable (FV) consumption will be assessed using dermal reflectance spectrometry (Veggie Meter, Longevity Link Corp). Carotenoids are red, orange, and yellow fat-soluble pigments found in FV, and non-invasively measured dermal carotenoids are a valid and reliable proxy for intake of red, orange, yellow and dark green FV in adults and children. Per standard protocol under the direction of Nancy Moran, PhD (co-investigator) one finger from each child will be scanned using the Veggie Meter (Longevity Link Corp) to provide a linear score that represents dermal carotenoid intensity (0-850). Skin carotenoid levels can range from 0-850 with 3.9% standard deviation (SD). Two readings will be collected and if there is more than 33 units (1 SD based on normative data from manufacturer) difference, a third will be collected.
Activity | baseline (T1), 10-11 weeks after baseline (T2), and 24- weeks after baseline (T3)
  Accelerometers (GT3X+ Actigraph, Pensacola, FL). Following standard protocols for young children41,84,111,112, toddlers will wear the activity monitors for 8-consecutive days with the goal of obtaining at least 4 days of valid wear time. We had increased compliance with wear time by providing CareAline wraps to the families in our pilot study. These wraps are stretchy Velcro-fastened covers that are usually used to protect central line ports from toddlers' curious hands. Research staff will show parents directly how to place the actigraph on their child. Parents will receive an instruction guide to take home for reference and they will be encouraged to call research staff if they have any questions about it at home. Parents will be instructed to keep a detailed log of the child's activity when the child wears the actigraph to differential low count data (sleep vs non wear vs sedentary). Parents will be instructed to return the actigraph during the next measurement session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be collected include toddler's anthropometric data, skin carotenoid levels, diet (parent report food frequency questionnaire), activity measured via wearable device, demographic qualities (parent report), food insecurity (parent report), and toddler temperament (parent report); parent's behaviors (self-report and observation) and perceptions of interventions (self-report). Data will be collected on parent-toddler dyads at three time points. To facilitate the interpretation and reuse of the data, a README file and data dictionary will be generated and deposited into a repository along with all shared datasets. The README file will include a description of data collection methods. The data dictionary will define and describe all variables in the dataset.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available as soon as possible but no later than within one year of the completion of the funded project period or upon acceptance of specific data for publication. Data will be available a minimum of 10 years after the completion of the funded project.
Access Criteria: Deidentified data will be made available as public use data to the research community via openIPSR. Users of the public use data must register with ICPSR and agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads.